CLINICAL TRIAL: NCT06755866
Title: DCE-MRI Based on 4D Free Breathing for Predicting Preoperative Neoadjuvant Chemoradiotherapy for Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLX2024-273
Record Dates: First submitted 2024-12-15; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application of DCE-MRI based on 4D Free Breathing in predicting the efficacy of preoperative neoadju (Experimental): Prospective collection uses a Philips 3.0T MRI scanner equipped with a dStream Torso 32-channel coil. DCE-MRI was performed using a free respiration sequence with a flow rate of 3.0 m/s. The medical images and clinical data related to esophageal cancer using 4D Free Breathing DCE-MRI technology were performed by two radiologists (one with 3 years of diagnostic experience and the other with 15 years of diagnostic experience), including subjective and objective assessment of image quality in the diagnosis of esophageal cancer, and the use of this technology to predict the efficacy of preoperative neoadjuvant chemoradiotherapy for esophageal cancer with pathological PCR as the outcome.
  Interventions: Diagnostic Test: The application value of MRI 4D Free Breathing DCE-MRI in the treatment of esophageal cancer

INTERVENTIONS:
Diagnostic Test: The application value of MRI 4D Free Breathing DCE-MRI in the treatment of esophageal cancer — Chest MRI scan outside of standard treatment options

SUMMARY:
To prospectively collect medical images and clinical data related to esophageal cancer using 4D Free Breathing DCE-MRI technology, to evaluate the image quality in the diagnosis of esophageal cancer, and to predict the efficacy of preoperative neoadjuvant chemoradiotherapy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age and older;
2. First diagnosis of esophageal squamous cell carcinoma confirmed by histopathological biopsy;
3. The clinical stage is cT1b~cT2N+; or the clinical stage is cT3~cT4 any N, (thoracic esophageal cancer, esophagogastric junction cancer);
4. There are no contraindications to MRI examination

Exclusion Criteria:

1. Have other primary tumors;
2. The image quality does not meet the diagnostic criteria;
3. Those who do not cooperate with the inspection;
4. Patients who have received prior chemoradiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response assessment | Surgery was performed within one month after neoadjuvant therapy, and the pathological pCR of the pathological results obtained from the surgery was used as the gold standard in this study to evaluate tumor treatment response
  This study aims to assess tumor treatment response using pathology gold standard pCR . pCR refers to the state in which the pathological tumor completely disappears after systemic therapy, such as chemotherapy, targeted therapy, or endocrine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China